CLINICAL TRIAL: NCT01806558
Title: Pilot Study: Combined Molecular Breast Imaging/Ultrasound System for Diagnostic Evaluation of MBI-detected Lesions
Acronym: MBI/US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-004900
Record Dates: First submitted 2013-03-01; First posted 2013-03-07 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; molecular breast imaging; breast; breast lesion
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Women with lesion on MBI (Experimental): Women with lesion on MBI
  Interventions: Procedure: Molecular Breast Imaging

INTERVENTIONS:
Procedure: Molecular Breast Imaging — Molecular breast Imaging is a new nuclear medicine technique for imaging the breast. It uses small filed of view semiconductor-based gamma cameras that use Cadmium Zinc Telluride detectors. These have superior spatial and energy resolution to conventional sodium iodide detectors.
  Other Names: MBI

SUMMARY:
A combined molecular breast imaging / ultrasound system will enable coregistration of a functional abnormality seen on Molecular Breast Imaging (MBI) with the corresponding anatomical abnormality seen on ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* The pilot study will comprise 12 women age 40 and older who have at least one of the following inclusion criteria:

  1. Have a finding of a mass lesion on mammography or breast MRI (BIRADS 0, 4 or 5) that is >0.5 cm and < 2 cm in size and has had or will have additional workup with focused ultrasound.
  2. Have a finding of a mass lesion on ultrasound (BIRADS 0, 4 or 5) that is > 0.5 cm and < 2 cm in size.
  3. Have a positive finding on MBI that is < 2 cm in size and requires additional diagnostic workup with focused ultrasound.

Exclusion Criteria:

1. Are unable to understand and sign the consent form
2. Are pregnant or lactating
3. Are physically unable to sit upright and still for 40 minutes
4. Have undergone bilateral mastectomy
5. Are not scheduled to undergo conventional ultrasound

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the potential benefits of co-registered MBI and ultrasonic information relative to independent acquisition of each modality. | 1 year
  Presence / absence of correlation between lesion seen on ultrasound and lesion seen on MBI.

CONTACTS AND LOCATIONS:
Overall Officials: Michael K O'Connor, PhD, R-D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Rhodes DJ, Hruska CB, Phillips SW, Whaley DH, O'Connor MK. Dedicated dual-head gamma imaging for breast cancer screening in women with mammographically dense breasts. Radiology. 2011 Jan;258(1):106-18. doi: 10.1148/radiol.10100625. Epub 2010 Nov 2. PMID 21045179
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0